CLINICAL TRIAL: NCT02461550
Title: Irreversible Electroporation Ablation for Colorectal Metastases to the Lung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-001
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2017-02

CONDITIONS: Colorectal Metastases to the Lung
Keywords: Irreversible Electroporation Ablation; 15-001
MeSH Terms: interventions — Electroporation

ARMS (1):
- IRE procedure (Experimental): The IRE procedure will be performed in the operating room at the time of scheduled clinical resection of colorectal lung metastases by the surgeon with guidance from the Interventional Radiologist.
  Interventions: Device: Irreversible Electroporation Ablation

INTERVENTIONS:
Device: Irreversible Electroporation Ablation

SUMMARY:
The investigators are investigating the use of a new cancer treatment called Irreversible Electroporation (IRE). This treatment delivers electrical energy between two needles placed in a cancer. The electrical energy causes cells to die. While this has been used in patients for different applications, the investigators are trying to understand how safe and well it works in colon cancer that has spread to the lung. Once the irreversible electroporation procedure is completed during the operation, the surgeon will then remove the cancer according to standard procedure. As part of the study, they will be measuring safety of the electrical energy delivered and will be reviewing the resected specimen under the microscope.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Colorectal cancer with oligometastatic colorectal cancer in the lung
* Lung lesion size is greater than 1 cm
* Patient will undergo surgical resection as per consultation with their thoracic surgeon and medical oncologist
* Patient is cleared to undergo paralytic anesthesia.
* Patients 18 years old and older

Exclusion Criteria:

* Patients with history of cardiac dysrhythmia
* Known heart failure (EF < 40%)
* Pacemaker/defibrillator
* Patient's with any metallic cardiac implant
* Patient on anti-coagulation therapy and are unable to stop therapy for the perioperative period
* Women who are pregnant and/or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Solomon, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- IRE Procedure: The IRE procedure will be performed in the operating room at the time of scheduled clinical resection of colorectal lung metastases by the surgeon with guidance from the Interventional Radiologist.
  Irreversible Electroporation Ablation
Period: Overall Study
Arm/Group | IRE Procedure
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IRE Procedure
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 42 [35 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: The Frequency of Adverse Events
Description: Safety will be measured by using the NCI Common Terminology Criteria for Adverse Events (CTCAE v4.0). The goal of this study is to establish safety.
  If there are 3 or more grade 3 or higher device related AEs, then we will stop the study.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | IRE Procedure
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | IRE Procedure
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IRE Procedure (N=2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Resp, thoracic & mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT02461550/Prot_SAP_000.pdf